CLINICAL TRIAL: NCT07325045
Title: Biomechanical Parameter Quantification and Finite Element Simulation of Lever Positioning Manipulation in Patients With Thoracolumbar Scoliosis
Brief Title: Biomechanical Study of Lever Positioning Manipulation on Scoliosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Tian Yv, Principal Investigator, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSLL-KY-2025-101-01
Record Dates: First submitted 2025-11-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lever positioning manipulation group (Experimental)
  Interventions: Procedure: Lever positioning manipulation

INTERVENTIONS:
Procedure: Lever positioning manipulation — 1 The patient took the prone position, exposed the waist and back, relaxed the whole body, and straightened the lower limbs. 2 The surgeon determined the top vertebra of the scoliosis according to the whole spine X-ray film, and used the olecranon of the elbow as the force fulcrum to accurately press the transverse process or spinous process on the convex side of the top vertebra, and the assistant fixed the shoulder of the patient. 3 The patient was asked to open his mouth and exhale, and the operator lifted the patient 's lower limbs on the other hand. Through the force arm conduction of the lower limbs-pelvis-spine, the lower limbs were lifted obliquely above the convex side to form a force arm lever. 4 When pulling to the resistance point, the surgeon pulled quickly with inch force. After the operation, the patient was allowed to rest in a prone position for 10 minutes.

SUMMARY:
Research background Scoliosis is a common three-dimensional spinal deformity, especially in adolescents. In severe cases, it can lead to thoracic deformation and cardiopulmonary dysfunction. At present, clinical treatment is mainly based on Cobb angle to take observation, brace or surgical intervention, but there are problems such as poor compliance and large trauma. As a non-invasive massage therapy, leverage positioning manipulation has shown orthopedic effects in clinical practice, but its biomechanical mechanism has not been systematically quantified, which restricts its standardization and promotion.

Purpose of the study The purpose of this study is to quantify the mechanical and kinematic parameters of lever positioning manipulation in the treatment of scoliosis through biomechanical testing and finite element simulation technology, to construct an individualized finite element model, to analyze the stress and strain distribution of each structure of the spine under the intervention of manipulation, to reveal its biomechanical mechanism, and to provide scientific basis for the standardization of manipulation and the optimization of curative effect.

Research contents and methods The study is divided into two parts : In the first part, 30 patients with scoliosis were recruited. Through the integrated mechanical sensor and motion capture system, the mechanical parameters ( such as preload force, maximum pull force ) and kinematic parameters ( such as angle, angular velocity ) during the manipulation were recorded in real time. In the second part, based on the CT data of patients, the three-dimensional finite element model of T10-L2 segment was constructed by using Mimics, Geomagic, SolidWorks and ANSYS software to simulate the loading process of manipulation and analyze the stress and strain response of vertebral body, intervertebral disc and ligament complex under the action of manipulation.

Expected results and significance This study will systematically quantify the biomechanical characteristics of lever positioning manipulation for the first time, and clarify its mechanism of action in the treatment of thoracolumbar scoliosis. Through the finite element simulation, the stress distribution is visualized, which provides data support for the precision and individualization of manipulation, promotes the transformation of massage manipulation from ' experience dependence ' to ' quantitative science ', and lays a theoretical foundation for the development of intelligent orthopedic equipment in the future.

Ethics and quality control The study has passed the ethical review, and all participants will sign the informed consent. The manipulation was performed by the same experienced physician, and the data collection and analysis process was strictly controlled to ensure that the results were true and reliable.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 and 45 years, stable vital signs, no severe diseases in other systems;
2. Diagnosed with scoliosis via standard anterior-posterior and lateral spinal radiographs, with a Cobb angle of 10° < θ <= 45°, and no severe complications;
3. No history of spinal surgery;
4. Voluntarily willing to participate in this study as a subject to undergo LPM procedures, and signing the informed consent form by themselves or their guardian. Note: Only patients meeting all of the above four criteria can be included in this study.

Exclusion Criteria:

1. Individuals with severe osteoporosis, spinal fractures, tumors, infections, or lesions within the spinal canal;
2. Those with related complications, such as cardiopulmonary insufficiency (NYHA class >= II) or severe neurological disorders;
3. Those with compression fractures or spinal cord injuries;
4. Individuals with cognitive impairment or mental disorders who cannot cooperate with biomechanical testing;
5. Those with a history of spinal surgery;
6. Those with severe skin lesions or dermatological diseases at the operation site;
7. Women who are menstruating, pregnant, planning pregnancy, or in the postpartum period;
8. Those with other conditions that may reduce the likelihood of completing the procedure, such as a fear of manual therapy;
9. Individuals with unclear surface markers, affecting motion capture accuracy (e.g., BMI >= 35 kg/m^2).

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
elbow pulling the maximum force：Through the mechanical gloves and elbow sleeves, the mechanical parameters in the process of manual operation were collected. | 2 weeks
  The operator wears mechanical measurement gloves and elbow sleeves to perform manual operation on the recipient. The mechanical parameters were collected by a pressure sensor, and the unit of measurement was Force ( Newton, N ). The average or peak value of each parameter was reported.

SECONDARY OUTCOMES:
maximum force of both hands pulling：Through the mechanical gloves and elbow sleeves, the mechanical parameters in the process of manual operation were collected. | 2 weeks
  The operator wears mechanical measurement gloves and elbow sleeves to perform manual operation on the recipient. The mechanical parameters were collected by a pressure sensor, and the unit of measurement was Force ( Newton, N ). The average or peak value of each parameter was reported.
lateral flexion angle： Through the three-dimensional motion capture system, the kinematic parameters of spinal activity during manipulation were collected. | 2 weeks
  The operator performs manual operation on the subject, and collects the kinematic parameters of the manual operation through the three-dimensional motion capture system equipment, and the measurement unit is : degree.
rotation angle： Through the three-dimensional motion capture system, the kinematic parameters of spinal activity during manipulation were collected. | 2 weeks
  The operator performs manual operation on the subject, and collects the kinematic parameters of the manual operation through the three-dimensional motion capture system equipment, and the measurement unit is : degree.
pulling time：Through the three-dimensional motion capture system, the time of the manipulation process is recorded. | 2 weeks
  The operator performs the manual operation on the subject, collects the kinematic parameters of the manual operation through the three-dimensional motion capture system equipment, and records the manual operation time at the same time. The measurement unit is seconds ( S ).
pulling angular acceleration：Through the three-dimensional motion capture system, the kinematic parameters of spinal activity during manipulation were collected. | 2 weeks
  The operator performs the manual operation on the subject, collects the kinematic parameters of the manual operation through the three-dimensional motion capture system equipment, and records the manual operation time and angular velocity. The acceleration is calculated and the average and maximum values are recorded.
extension angle：Through the three-dimensional motion capture system, the kinematic parameters of spinal activity during manipulation were collected. | 2 weeks
  The operator performs manipulation on the subject, collects the kinematics parameters of the manipulation through the three-dimensional motion capture system equipment, and records the angle.
preloading force of both hands：Through the mechanical gloves and elbow sleeves, the mechanical parameters in the process of manual operation were collected. | 2 weeks
  The operator wears mechanical measurement gloves and elbow sleeves to perform manual operation on the recipient. The mechanical parameters were collected by a pressure sensor, and the unit of measurement was Force ( Newton, N ). The average or peak value of each parameter was reported.
Elbow preload force：Through the mechanical gloves and elbow sleeves, the mechanical parameters in the process of manual operation were collected. | 2 weeks
  The operator wears mechanical measurement gloves and elbow sleeves to perform manual operation on the recipient. The mechanical parameters were collected by a pressure sensor, and the unit of measurement was Force ( Newton, N ). The average or peak value of each parameter was reported.
average pulling angular velocity：Through the three-dimensional motion capture system, the kinematic parameters of spinal activity during manipulation were collected. | 2 weeks
  The operator performs manipulation on the subject. The kinematics parameters of the manipulation are collected by the three-dimensional motion capture system equipment, the angle change and time are recorded, the angular velocity is calculated, and the average value and the highest value are calculated.
The stress of each structure：Through the analysis of finite element software, the stress of the spine under the intervention of manipulation was simulated. | 2 weeks
  The kinematics and mechanics data of the manipulation operation measured above were statistically analyzed. These data were input into the three-dimensional finite element model of the spine to simulate the manipulation. Through the finite element software analysis, the stress change cloud map and data of the spine were obtained, including the average value and the maximum and minimum values.
Strain of each structure：Through the analysis of finite element software, the strain of the spine under the intervention of manipulation was simulated. | 2 weeks
  The kinematics and mechanics data of the manipulation of the previous measurement were statistically analyzed. The data were input into the three-dimensional finite element model of the spine to simulate the manipulation. Through the analysis of the finite element software, the strain cloud map and displacement data of the spine were obtained, including the average value and the maximum and minimum values.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No